CLINICAL TRIAL: NCT02855008
Title: Steps to Effective Problem Solving in Group Homes for Individuals With Intellectual Disabilities
Brief Title: Steps to Effective Problem Solving in Group Homes
Acronym: STEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sarah Ailey, Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD086211 (NIH); 1R01HD086211-01A1 (NIH)
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Problem Behavior
Keywords: Social Problem-Solving; Intellectual Disability; Problem Behaviors; Community based intervention; Prevention
MeSH Terms: conditions — Problem Behavior; Intellectual Disability | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STEPS (Experimental): Experimental: Individuals with ID and residential staff in group homes receive 6 one-hour STEPS sessions over 12 weeks and a booster in week 18 following a standardized manual. Sessions include interactive games to build group cohesiveness, along with interactive discussion and practice. Participants are given session materials and 1-2 worksheets to practice learned skills and are asked to return the worksheets at the next session. Residential staff are given additional materials with tips on how to help residents practice social problem-solving skills between sessions. Highlights of each session using a standardized format are brought to the following session to help with engagement and provide cues for retention of materials.
  Interventions: Behavioral: STEPS
- Food for Life (Active Comparator): Active Comparator: Individuals with ID and residential staff in group homes receive 6 one-hour Food for Life sessions over 12 weeks and a booster in week 18 following a standardized manual. Sessions include interactive games regarding food and nutrition followed, along with interactive discussion and practice. Participants are given session materials and 1-2 worksheets to practice learned skills and are asked to return the worksheets at the next session. Residential staff are given additional materials with tips on how to help residents practice Food for Life skills between sessions. Highlights of each session using a standardized format are brought to the following session to help with engagement and provide cues for retention of materials.
  Interventions: Behavioral: Food for Life

INTERVENTIONS:
Behavioral: STEPS — Agencies providing residential services to individuals with ID gave us letters of agreement (N=9) when we submitted for funding. We randomized these agencies and followed the specific order. Over the past year, recruitment issues have resulted in our only being able to recruit at six of the original nine agencies. To address the issues, we compiled a list of 15 additional local agencies within a 50 mile radius. We are recruiting from an additional six agencies and are in contact with another four. We also changed our recruitment criteria to include co-ed homes. Within each agency we then, (1) determine homes that that meet criteria and, by gender (male, female, co-ed), randomize to STEPS or attention-control condition. Residential staff are consented first. Individuals with ID (or guardians if they have one) are then consented. 18 homes will participate in STEPS.
  Arms: STEPS
Behavioral: Food for Life — Agencies providing residential services to individuals with ID gave us letters of agreement (N=9) when we submitted for funding. We randomized these agencies and followed the specific order. Over the past year, recruitment issues have resulted in our only being able to recruit at six of the original nine agencies. To address the issues, we compiled a list of 15 additional local agencies within a 50 mile radius We are recruiting from an additional six agencies and are in contact with another four. We also changed our recruitment criteria to include co-ed homes. Within each agency we then, (1) determine homes that that meet criteria and, by gender (male, female, co-ed), randomize to STEPS or attention-control condition. Individuals with ID and staff are recruited after randomization. Residential staff are consented first. Individuals with ID (or guardians if they have one) are then consented. 18 homes will participate in Food for Life.
  Arms: Food for Life

SUMMARY:
Aggressive/challenging behaviors in individuals with intellectual disability are a major public health concern for them, their families, their service programs and staff, and their communities. This randomized clinical trial will test the efficacy and cost effectiveness of a preventive community-based social problem solving intervention, the Steps to Effective Problem-solving (STEPS), delivered in group homes. The program uses residential staff participation and the group environment to facilitate improved social problem solving skills and reduce aggressive/challenging behaviors in this population in group homes and work settings.

DETAILED DESCRIPTION:
Aggressive/challenging behaviors (AC/Bs) are a major public health problem for individuals with intellectual disabilities (ID) living in group homes. A leading reason for psychiatric hospitalizations and incarcerations, A/CBs are costly to the healthcare system, agencies and families. Social problem solving (SPS) training programs for individuals with ID have had positive behavioral results, but most were conducted in clinical or forensic settings. None were community-based preventive interventions, none examined whether A/CBs decreased in participants' group homes and work settings, and none addressed cost effectiveness. In preliminary work, the investigators modified an effective SPS training program, using input from individuals with ID and residential staff, as a preventive intervention for the group home setting. Steps to Effective Problem-solving (STEPS) includes residential staff and uses the group home environment to facilitate behavior change. The purpose of this clinical trial is to test the efficacy of STEPS for individuals with ID. Specific aims are to 1) Assess the efficacy of the STEPS intervention in group homes to improve SPS skills and reduce A/CBs of the individuals with ID compared to an attention-control nutrition program from baseline to 12, 24 and 36 weeks, controlling for behavioral determinants of A/CBs (demographics, agency/home environment, current health). 2) Assess the mediating effect of the support environment for SPS (residential staff SPS skills, group home level SPS skills, and group cohesiveness) on the improvement of SPS skills and reductions in A/CBs. 3) Evaluate cost effectiveness of STEPS relative to usual care for A/CB incidents in group homes. The investigators expect to show STEPS to be a preventive behavioral strategy to reduce A/CBs among individuals with ID, improve the cost effectiveness of their care and make an important incremental advance in SPS research.

ELIGIBILITY:
Inclusion/exclusion criteria

Group home

Inclusion criteria:

* Serve individuals with mild to moderate ID;
* Have at least 10 A/CB incident reports in resident files over the prior six-month period, with at least 30% of residents in each home having incident reports in that period
* Have 4 or more residents, with a minimum of 3 agreeing to participate
* Individuals with ID and residential staff all speak English
* Have at least one residential staff members who agree to participate.

Exclusion criteria:

* If group home specifically serves individuals with ID who also have serious mental illness (e.g., severe autism, schizophrenia)
* If group home specifically serves forensic populations
* If the group home participated in previous preliminary study

Individual with ID

Inclusion criteria:

* Has mild to moderate ID (operationalized as IQ 50-75 per agency records) and mild to moderate limitations in adaptive functioning (measured by the Inventory for Client and Agency Planning used in all residential agencies in Illinois, per agency record)
* Lives in a chosen group home
* Is verbal and speaks English

Exclusion Criteria:

* If individual does not meet inclusion criteria and
* If participated in the preliminary study

Residential staff

Inclusion criteria:

* Employed as residential staff in the chosen group homes and
* Speak and read English

Exclusion criteria:

* Does not meet inclusion criteria
* Participated in the previous preliminary study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The Iowa Family Interactions Rating Scales (IFIRS) Individual-level Problem-solving scales | Baseline, 12, and 24 weeks
  Change from baseline Individual with ID SPS: Uses a 15-20 minute videotape of a problem-solving interaction of the group of individuals with ID living in the group home and their residential staff to assess individuals with ID SPS skills - solution quantity, solution quality, effective process, disruptive process, and negotiation/compromise at the individual level.
Problem-solving Task (PST) | Baseline, 12, and 24 weeks
  Change from baseline Individual with ID SPS: Has four questions on each of five problem vignettes that measure individual with ID SPS skills. The vignettes are read by data collectors to the individuals and responses audiotaped.
The IFIRS Dyadic-interaction scales | Baseline, 12 and 24 weeks
  Change from baseline Individual with ID Behaviors: Uses the same 15-20 minute videotape of a problem-solving interaction to assess individual with ID A/CBs. Items include hostility, verbal attack, physical attack, contempt, etc. (total 22 items) of each individual with ID
General Maladaptive Index | Baseline, 12 and 24 weeks
  Change from baseline Individual with ID Behaviors: Qualified Intellectual Disability Professionals (QIDPs) at the residential agency and work setting supervisors (sheltered workshops and employment) will be asked to fill out the GMI on participants with ID. The GMI measures the frequency (0 = never to 5 = one or more times an hour) and severity (0 = not serious to 4 = extremely serious) of problem behaviors in eight domains (hurtful to self or others, destructive, disruptive, socially offensive, unusual/repetitive, withdrawn/inattentive, uncooperative).
Agency incident reports | For 24 weeks prior to intervention, 12, 24 and 36 weeks
  Change from baseline Individual with ID behaviors: Residential staff members fill out incident reports. The reports are reviewed by QIDPs, kept in resident files, and tracked by the agencies. Data will be abstracted from agency tracking records and de-identified. The investigators will analyze counts of incidents for outcomes and summarize descriptive data of key elements of the incident reports.

SECONDARY OUTCOMES:
The Iowa Family Interactions Rating Scales (IFIRS) Individual-level Problem-solving scales | Baseline,12 and 24 weeks
  Change from baseline Residential staff SPS (Support environment for Individual with ID). Uses the same 15-20 minute videotape of a problem-solving interaction of the group of individuals with ID living in the group home and their residential staff to assess residential staff SPS skills - solution quantity, solution quality, effective process, disruptive process, and negotiation/compromise at the individual level.
Social Problem Solving Inventory Revised - Short form (SPSI-R SF) | Baseline, 12 and 24 weeks
  Change from baseline Residential staff SPS (Support environment for Individual with ID). The five dimensions of this measure are positive attitude, negative attitude, rational style, impulsive/careless style, and avoidant style.
IFIRS Group Problem-solving Scales | Baseline,12 and 24 weeks
  Change from baseline of Group (of individuals with ID and their residential staff) SPS (Support environment for Individual with ID). The scales include problem-solving enjoyment, agreement on problem description/solution, implementation, and problem difficulty for group,
Group Environment for the Intervention Scale (GEIS) | Week 1 and 12
  Change from baseline of group environment - cohesiveness (Support environment of individual with ID). The GEIS is a 25-item measure of group environments. The three subscales are implementation and preparedness, counter-productive activity, and cohesiveness. The GEIS will be scored using audiotapes from Sessions 1 and 6 by trained research assistants.

OTHER OUTCOMES:
Life events section of Psychiatric Assessment Schedule for Adults with Developmental Disabilities | Baseline, 12 and 24 weeks
  Change from baseline in A/CB determinant of life events: (17 items 2-recent 1-event 0-never)
Glasgow Depression Scale for People with Learning Disabilities [GDS-LD]) | Baseline, 12 and 24 weeks
  Change from baseline of A/CB determinant depression. The GDS-LD was developed for use among individuals with ID (called "learning disabilities" in the UK). It has a sensitivity ranging from 90-96% and specificity ranging from 83.9-90%, with a score of 13.
Medication management | Baseline, 12 and 24 weeks
  Background information on psychotropic medications will be gathered from agency records
A/CB incident costs | 12-36 weeks
  Compare A/CB incident costs for experimental arm vs. active comparator arm. The investigators will evaluate the cost-effectiveness of STEPS from the societal perspective, taking into account costs borne by the program, group home, health care system, public services, participant, and family. The STEPS experimental arm group will be compared to usual care (active comparator Food for Life) group costs of A/CBs excluding costs of the nutrition intervention). We will calculate the net cost (or net savings) associated with STEPS vs. Food for Life arms, such that the net cost = program-related cost - A/CB incident cost

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H Ailey, PhD RN, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share aggregated data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and informed consent can be shared now. Expect to share preliminary results Fall '22
Access Criteria: Other researchers

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT02855008/Prot_SAP_002.pdf
  • Informed Consent Form (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT02855008/ICF_003.pdf